CLINICAL TRIAL: NCT02450721
Title: Clinical and Laboratory Biomarkers in Patients With Atherothrombotic Stroke
Acronym: CLAST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: St. Petersburg State Pavlov Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: StPetersburgSPMU
Record Dates: First submitted 2015-05-19; First posted 2015-05-21 (Estimated); Last update posted 2016-05-04 (Estimated); Status verified 2016-05

CONDITIONS: Carotid Artery Diseases; Stroke
Keywords: atherosclerosis; biomarkers; carotid artery stenosis; ischemic stroke.
MeSH Terms: conditions — Carotid Artery Diseases; Stroke; Atherosclerosis; Carotid Stenosis; Ischemic Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Acute stroke: Patients in the acute phase of atherothrombotic stroke or TIAs with 50-99% ACAS within the first 3 days af vascular event.
  Interventions to be administered: Biomarkers serum level measurement, history taking, neurological examination, duplex ultrasound, MMSE, National Institutes of Health Stroke Scale (NIHSS)
  Interventions: Other: Biomarkers serum level measurement
- Stable carotid artery stenosis: Patients with 50-99% ACAS without history of vascular events during one month before enrollment.
  Interventions to be administered: Biomarkers serum level measurement, history taking, neurological examination, duplex ultrasound, MMSE
  Interventions: Other: Biomarkers serum level measurement
- Control group: Healthy volunteers without ACAS Interventions to be administered:Biomarkers serum level measurement, history taking, neurological examination, duplex ultrasound, MMSE
  Interventions: Other: Biomarkers serum level measurement

INTERVENTIONS:
Other: Biomarkers serum level measurement — Biomarker serum level measurement was performed with ELISA using following kits: Lp-PL-A2 ELISA- "Cloud-CloneCorp." (USA); PAPP-A ELISA- "IBL" (Germany); Lp (a) ELISA Kit-"AssayPro" (USA ), ADMA ELISA Kit- "ImmunDiagnostik" ( Germany); hsCRP ELISA- "Biomerica" (Germany); according to the manufacturer's instructions . Absorbance of standards and samples was measured with a microplate reader "Bio-Tek" (USA) at a wavelength specified by the kit manufacturer . The calculation of the determined biomarkers concentration was performed using the software SOFTmaxPRO.

SUMMARY:
Aim of the present study is to investigate molecular and clinical markers in patients with atherosclerotic carotid stenosis (ACAS) in the ischemic stroke acute phase.

DETAILED DESCRIPTION:
Background: Laboratory biomarkers of atherosclerosis can be valuable in decision about operative treatment in patients with mild to severe atherosclerotic carotid stenosis (ACAS) and high stroke risk. However nowadays there are no established instruments for personalized atherothrombotic stroke diagnostics. Aim of the present study was to access atherosclerosis biomarkers serum levels in patients with ACAS during the ischemic stroke/ transient ischemic attack (TIA) acute phase.

Main objective of the study To explore informative biomarkers to determine the risk of stroke in patients with significant ACAS.

Secondary objectives

1. To investigate the association between the degree of neurological and cognitive deficits , the features of the disease , the severity of brain lesions according to neuroimaging data with the concentration of lipoprotein -associated phospholipase A2 (LP-PL-A2), high sensitive C- reactive protein (hsCRP) , pregnancy-associated plasma protein A (PAPP-A), asymmetric dimethylarginine (ADMA), lipoprotein (a) in patients with atherothrombotic stroke.
2. To find the most valuable laboratory biomarkers of atherosclerosis , to compare them with clinical and objective data to make decision about inclusion of these biomarkers in routine practice as a screening test of atherosclerotic plaque instability and for stroke risk prediction and in decision about operative treatment in patients with ACAS.

Design and Methods A single-blind cross-sectional trial was performed to investigate laboratory biomarkers of atherosclerosis in patients with atherosclerotic stenosis of the internal carotid artery 50-99 % , and in healthy volunteers. Randomizing and blinding technique: laboratory scientist and statistician do not have information about the belonging of biomaterials patient to any of the groups studied .

Examination of patients includes history taking, neurological examination, duplex ultrasound, mini mental score examination (MMSE), enzyme-linked immunosorbent assay (ELISA) performed atherosclerosis biomarkers serum level measurement (LP-PL-A2, PAPP-A, ADMA, hsCRP and blood lipid profile).

ELIGIBILITY:
Acute stroke

Inclusion Criteria:

* 50-99% atherosclerotic carotid artery stenosis
* Acute atherothrombotic stroke/TIA (according to TOAST-criteria) within the first 3 days after vascular event

Exclusion Criteria:

* risk factors of non-atherothrombotic stroke (according to TOAST-criteria)
* cancer
* exacerbation of decompensated chronic diseases
* infections
* acute cardiovascular diseases
* large operation during 1 month before enrollment
* Cortexin, Actovegin, Cerebrolysin, Erythropoetin administration during 1 week before enrollment.

Stable ACAS

Inclusion Criteria:

* 50-99% atherosclerotic carotid artery stenosis
* no history of vascular events during one month before enrollment

Exclusion Criteria:

* risk factors of non-atherothrombotic stroke (according to TOAST-criteria)
* cancer
* exacerbation of decompensated chronic diseases
* infections
* acute cardiovascular diseases
* large operation during 1 month before enrollment
* Cortexin, Actovegin, Cerebrolysin, Erythropoetin administration during 1 week before enrollment.

Control group

Inclusion Criteria:

* intima media thickness less then 1mm
* no history of stroke/TIAs

Exclusion Criteria:

* risk factors of non-atherothrombotic stroke (according to TOAST-criteria)
* cancer
* exacerbation of decompensated chronic diseases
* infections
* acute cardiovascular diseases
* large operation during 1 month before enrollment
* Cortexin, Actovegin, Cerebrolysin, Erythropoetin administration during 1 week before enrollment.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In-hospital patients
Sampling Method: Non-Probability Sample
Enrollment: 97 (Estimated)
Dates: Start 2011-01; Primary Completion 2015-01 (Actual); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Mean concentration of Lipoprotein-associated Phospholipase A2 (LP-PL-A2) | 0 month
Mean concentration of Pregnancy-associated Plasma Protein A (PAPP A) | 0 month
Mean concentration of Asymmetric Dimethylarginine (ADMA) | 0 month
Mean concentration of highsensitivity C-reactive Protein (hsCRP) | 0 month
Mean concentration of Lipprotein (a) | 0 month

CONTACTS AND LOCATIONS:
Locations (1):
- StPetersburgSPMU, Saint Petersburg, Sankt-Peterburg, Russia